CLINICAL TRIAL: NCT06040801
Title: Effect of Geriatric Intervention in Frail Patients with Gastric, Biliary, and Pancreatic Cancer Receiving Palliative Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202002181B0A3; CMRPG3L1611 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2023-08-29; First posted 2023-09-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: GI Cancer
Keywords: Frailty; Comprehensive Geriatric Assessment (CGA); Chemotherapy; Outcome
MeSH Terms: conditions — Gastrointestinal Neoplasms; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frail group (Experimental): All patients receive a frailty assessment within 7 days before initiating the first cycle of palliative chemotherapy, followed by geriatric intervention. Patients exhibiting impairments in at least two dimensions are considered frail. The frail group will receive management and recommendations based on the specific impairment domain.
  Interventions: Behavioral: Frailty intervention measures
- Non-frail group (No Intervention): All patients receive a frailty assessment within 7 days before initiating the first cycle of palliative chemotherapy, followed by geriatric intervention. Patients exhibiting impairments in at least two dimensions are considered frail. The non-frail group will not receive additional interventions, but the clinical physicians will still provide appropriate treatment based on the patient's condition.

INTERVENTIONS:
Behavioral: Frailty intervention measures — Providing management and recommendations based on the specific impairment domain.
  Assessment domain:
  * Functional status
  * Nutrition
  * Comorbidity
  * Mobility/Falls
  * Mood
  * Cognition
  * Polypharmacy
  * Social support.
  Arms: Frail group

SUMMARY:
Gastric, biliary and pancreatic cancer are commonly malignancies from gastro- intestinal tract in Taiwan. Because lack of specific symptoms at presentation and effective screening methodology, majority of these patients are diagnosed with metastatic or unresectable disease. Palliative chemotherapy is the good standard of therapy for patients with unresectable gastric, biliary and pancreatic cancer with benefit of prolong survival time and improve quality of life.

Although the benefit of palliative chemotherapy seems to be the same for elderly and young cancer patients in clinical study, elderly patients are less frequently treated with chemotherapy or treated with suboptimal dosage. Elderly patients do not receive palliative chemotherapy because concerns of elder age, comorbidity, poor performance, lack of social/economic support and worry about treatment toxicities.

The increase in life expectancy of the general population resulted in an increase in the number of elderly patients with cancers referred for palliative chemotherapy. Overtreatment may result in high mortality due to disregard of the aging patients' frailty; on the other hand, under-treatment resulting from over-concern regarding their ability to tolerate treatment, may compromise the survival outcome. Therefore, the appropriately selection of geriatric cancer patients for palliative chemotherapy has to be addressed urgently.

Frailty is a progressive decline of physiological reserve leading to multiple functional disability and increases vulnerability to subsequent morbidity and mortality. Frailty is associated with treatment toxicity, chemotherapy tolerance, and survival outcome in clinical oncology. Recent randomized study reported geriatric intervention significantly improved chemotherapy tolerance in elderly patients. Therefore, the American Cancer Association has recommended routine geriatric assessment and intervention in oncogeriatric patients upon providing antitumor treatments. However, the effect of geriatric intervention on chemotherapy tolerance is seldom in Taiwan.

This study is an open, randomized, prospective trial to evaluate the effect of geriatric intervention on chemotherapy tolerance in patients with unresectable gastric, biliary, and pancreatic cancer. All patients with receive frailty assessment within 7 days before initiation of first cycle palliative chemotherapy followed by geriatric intervention. The study aim is to compare for chemotherapy tolerance, treatment-related toxicity, and quality of life after completion 3 months chemotherapy treatment course between frail and non-frail patients. This study also aims to explore the effect of geriatric intervention of treatment tolerance, treatment-related toxicity, and quality of life in frail patients with gastric, biliary, and pancreatic cancer receiving palliative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged sixty-five or older with metastatic or unresectable gastric, biliary, and pancreatic cancer.
* The patient must sign the informed consent form.
* Estimated survival period of more than 3 months.
* Conscious and able to communicate verbally or in writing, and willing to cooperate with invasive procedures.

Exclusion Criteria:

* Patients with cognitive impairment or unable to cooperate with the interventional procedures as determined by the clinical physician.
* Patients receiving concurrent other anticancer treatments (radiation or surgery).
* Patients with multiple types of cancer requiring simultaneous treatment.
* Patients who have previously participated in this study during a prior chemotherapy regimen.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Examine the completion rate of chemotherapy in frail and non-frail patient groups three months after treatment initiation to assess whether frailty affects tolerance. | After completion 3 months chemotherapy treatment.
Utilize CTCAE v5.0 to assess the grade and frequency of adverse events and treatment-related toxicity in frail and non-frail patient groups, and compare the differences between the two. | After completion 3 months chemotherapy treatment.
Assess the level of quality of life in frail and non-frail patient groups before and after treatment using EORTC QLQ-C30 v3 and EORTC QLQ-ELD14. | After completion 3 months chemotherapy treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan